CLINICAL TRIAL: NCT02383784
Title: Effects of Low- or High-glycemic Index Diets in Metabolic and Inflammatory Responses in Type 2 Diabetics
Brief Title: Effects of Low- or High-glycemic Index Diets on Metabolic and Inflammatory Responses in Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Vicosa (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Dr Junia Maria Geraldo Gomes, MSc, Federal University of Vicosa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 40501156099
Record Dates: First submitted 2015-02-26; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-GI diet (Experimental): Low glycemic index diet
  Interventions: Dietary Supplement: Low GI index diet
- High-GI diet (Experimental): High glycemic index diet
  Interventions: Dietary Supplement: High GI diet

INTERVENTIONS:
Dietary Supplement: Low GI index diet — Low glycemic index diet
  Arms: Low-GI diet
Dietary Supplement: High GI diet — High glycemic index diet
  Arms: High-GI diet

SUMMARY:
Background/Aims: Verify the effects of glycemic index (GI) on body composition, and on inflammatory and metabolic markers concentrations. Methods: Eighteen type 2 diabetics, (aged 42.4 + 5.1 years, BMI 29.2 + 4.8 kg.m-2) were randomly allocated to low GI (LGI) or high GI (HGI) groups. High or low GI meals were provided in the laboratory twice a day during 30 consecutive days. The other meals were consumed under free living condition and subjects were instructed to select foods presenting GI values corresponding to the allocated group. Body composition (body mass index, body fat percentage, waist circumference and waist-hip ratio), and inflammatory markers concentrations (interleukin-6, tumor necrosis factor-alpha, high molecular weight adiponectin, ultra-sensitive C-reactive protein and fibrinogen) and metabolic markers (glucose, insulin, total cholesterol, HDL cholesterol, free fatty acids, triglycerides and fructosamine) were assessed at baseline and after intervention. Food intake was monitored during the study. The criterion for statistical significance was P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Level of physical activity light to moderate
* Use of sulfonylureas or biguanides oral hypoglycemic drugs
* Stable medications for the previous 3 months

Exclusion Criteria:

* Cardiovascular, renal, or liver disease
* Treatment for cancer
* Smokers
* Daily consumption of > 50g/day of alcohol
* Pregnant, lactating, postmenopausal women,
* Hormone replacement therapy
* Recent change (last three months) in the level of physical activity or diet
* Weight instability (> 3 kg in the previous three months),
* Therapeutic diet
* Allergies, test foods intolerance
* Use of drugs affecting body metabolism and/or food intake.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-03; Primary Completion 2007-03 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Body fat content determined by tetrapolar bioelectrical impedance . | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Metabolism and body composition laboratory, Federal University of Vicosa, Viçosa, Minas Gerais, Brazil